CLINICAL TRIAL: NCT06331325
Title: Clinical Comparison of Frenotomy and Frenectomy Surgical Techniques for Management of High Frenum Attachment in Adult Patients: A Randomized Clinical Trial
Brief Title: Comparison of Frenotomy and Frenectomy Techniques for Management of High Frenum Attachment in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Nada Zazou, Lecturer of Periodontology, October University for Modern Sciences and Arts
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 724
Record Dates: First submitted 2024-03-20; First posted 2024-03-26 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: High Frenum Attachment
Keywords: frenum, labial; frenectomy
MeSH Terms: interventions — Oral Frenectomy

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial. Allocation Ratio: 1:1
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors will be unaware of the recruitment group. The allocation sequence will be contained within sequentially numbered, opaque, sealed packets that the patients will pull. According to the randomization table, the written number on the paper will allocate the patient to the intervention or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Frenotomy procedure (Experimental): Two C-shaped partial thickness incisions are performed on the two sides of the frenum leaving the underlying periosteum intact. Relocation of the muscle attachment is performed by blunt dissection using a mucoperiosteal elevator. Undermining or separation of the epithelium from the underlying lip mucosa is then performed by blunt dissection to facilitate tension-free suturing. The epithelium is then sutured to the underlying periosteum using three interrupted periosteal sutures and is left to heal by secondary intention.
  Interventions: Procedure: Frenotomy
- Frenectomy procedure (Active Comparator): Frenectomy group (Control): Two full-thickness incisions are performed apical and coronal to the frenum attachment and extending down to and including the periosteum. Complete excision of all muscle tissues is ensured and then both epithelial edges are approximated using single interrupted sutures achieving primary closure.
  Interventions: Procedure: Frenectomy

INTERVENTIONS:
Procedure: Frenotomy — Partial thickness procedure aiming to relocate high frenum attachment to a more apical level.
  Other Names: Frenal relocation
  Arms: Frenotomy procedure
Procedure: Frenectomy — Full-thickness excision of the frenum down to the bone level and suturing by achieving primary closure.
  Arms: Frenectomy procedure

SUMMARY:
The goal of this randomized clinical trial is to compare frenotomy to frenectomy surgical techniques in the management of high frenum attachment in adults. The main questions it aims to answer are:

* Does Frenotomy procedure have a lower relapse rate compared to frenectomy?
* Does Frenotomy procedure result in fewer postoperative complications? Participants will be divided into two groups. The intervention group will involve frenotomy procedure for participants and will be compared to the traditional frenectomy procedure in the comparator group. The level of the frenum will be measured at baseline and after 6 months. Pain scores will be recorded by the participants during the first week.

DETAILED DESCRIPTION:
Frenum is a triangular thin folded mucus membrane with underlying connective tissue and muscular fibers that attaches the lips and cheeks with alveolar mucosa enhancing the stability of the lip (Newman et al., 2020).

High frenum attachment can have numerous negative effects when highly attached close to the gingival margin including gingival recession, papilla loss, and obliteration of the sulcus, which might enhance plaque accumulation indirectly by hindering tooth brushing. It may also be responsible for midline diastema (Miller, 1985).

According to Mirko et al. (1974), there are four different types of labial frenal attachments: mucosal, gingival, papillary, and papilla piercing. The mucosal form is the most common and predominates in the mandible (Jańczuk & Banach, 1980).

Frenectomy procedure involves the complete removal of the frenum along with its attachment to the underlying bone. Frenotomy procedure is the incision and relocation of the frenal attachments to a more apical level (Dibart & Karima, 2008). However, this procedure is not well-documented in the literature and little is known about its expected relapse rates.

The rationale for conducting the research:

The traditional frenectomy procedure as described by Archer (1961) and Kruger (1964) could be considered invasive and may lead to scarring, delayed healing, and loss of the interdental papilla due to bone exposure and complete removal of fibers which may have negative esthetic outcome in addition to the frequent relapse rate (Devishree et al., 2012). A systematic review (Delli et al., 2013) discussed some complications that may arise when performing frenectomy procedure such as scar formation, postoperative pain, and swelling. Thus, frenectomy is considered a radical procedure with potential complications.

In contrast, frenotomy could be introduced as a more conservative procedure that can achieve the same outcomes with lower postoperative complications and scar formation. To the best of our knowledge, no studies are comparing both techniques in terms of relapse rate and postoperative pain.

Thus, the rationale of our study is to evaluate the clinical effectiveness of frenotomy procedure and its effect on frenum relapse and postoperative pain compared to the conventional frenectomy procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adults with active highly attached maxillary/mandibular labial frenum.
* Systemically healthy
* Non-smokers
* Gingival and plaque index <10%

Exclusion Criteria:

* Poor oral hygiene.
* Smokers
* Any systemic diseases or medications that delay wound healing.
* Pregnant or lactating females
* Previous frenal procedures.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Rebound / Relapse. | 6 months
  The level of the frenum will be measured at baseline and follow-up using William's graduated periodontal probe. The incisal edge will be assigned as a reference point at baseline to measure the frenum level before and after the procedure and identify the change in level.

SECONDARY OUTCOMES:
Postoperative pain | 1 week
  A visual analog scale (VAS) will be recorded by the patients during the first week postoperatively to compare the postoperative pain experienced after both procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Nada Zazou, PHD, Principal Investigator — Modern Sciences & Arts University
Locations (1):
- MSA University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, Statistical analysis.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data is available
Access Criteria: Shared upon request